CLINICAL TRIAL: NCT05078281
Title: Predictive Response Factors in Respondent Patients and Results After Monoplane Switch in Patients With Severe Eosinophilic Asthma Treated With Benralizumab
Brief Title: Patients With Severe Eosinophilic Asthma Treated With Benralizumab
Acronym: Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-BEN-2020-01
Record Dates: First submitted 2021-09-15; First posted 2021-10-14 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Asthma; Eosinophilic
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients with severe eosinophilic asthma receiving benralizumab.

SUMMARY:
Retrospective, multicenter, routine clinical practice study with consecutive inclusion of adult patients with severe eosinophilic asthma receiving benralizumab treatment.

DETAILED DESCRIPTION:
Retrospective study studying severe eosinophilic asthma. Patients with this disease who are on benralizumab treatment for at least 4 months before the start of the study will be included.

The purpose of this study is to analyze the predictive factors of response in patients with this type of disease treated with benralizumab, who obtain a complete response during their follow-up.

The results of the study will be obtained through the review of medical records, where demographic characteristics such as age, gender and smoking will be assessed; presence of comorbidities; clinical-functional variables; response variables (exercises, cycles of oral corticosteroids, admissions, visits to the emergency room or unscheduled, cumulative dose of oral corticosteroids, absenteeism from work) and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years of age) diagnosed with severe eosinophilic asthma on benralizumab treatment for at least 4 months from the start of the study.

Exclusion Criteria:

* Patients for whom no previous history is available or who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with severe eosinophilic asthma receiving benralizumab belonging to the health area of each center, in the Pulmonology and Allergology units, will be included. Patients must have at least 4 months of benralizumab treatment at the start of the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Response predictors in patients treated with benralicumab. | Up to 60 weeks.
  To analyze response predictors in patients with severe eosinophilic asthma under treatment with benralizumab who obtain a complete response during their follow-up.

SECONDARY OUTCOMES:
Study the response variables to benralizumab. | Up to 60 weeks.
  Number of visits to the emergency room or hospital admissions observed since the beginning of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gómez-Ballesteros Fernández, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain